CLINICAL TRIAL: NCT04434157
Title: Association of the Neutrophil/Lymphocyte Ratio and Lymphocyte /Platelet Ratio With Clinical Complications and Mortality in COVID-19 Patients
Brief Title: Association of the Neutrophil/Lymphocyte Ratio With Clinical Complications and Mortality in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Hospital Regional de Alta especialidad de Ixtapaluca (Other)
Collaborators: Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Omar Ramos-Peñafiel, Christian Ramos Peñafiel, MD, PhD, Hospital Regional de Alta especialidad de Ixtapaluca
Other Study IDs: NR-09-2020
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Covid-19
Keywords: Clinical Complications; Mortality Risk; COVID-19; Neutrophil/Lymphocyte Ratio
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is little information about the clinical characteristics and risk factors of Covid-19 in Latin American countries considering the ethnic differences and the high prevalence of obesity and cardiometabolic diseases. The aim of the study was to evaluate the association between laboratory tests and the risk of complications in SARS-CoV-2 infection and to determine their mortality risk factors in a sample of the Mexican population.

A retrospective cross-sectional study of the routinely collected data was performed in the Hospital Regional de Alta Especialidad de Ixtapaluca (HRAEI), State of Mexico. Adult patients (aged ≥18 years) with positive RT-PCR for SARS-CoV-2 and oxygen support that were admitted between March 28 and May 5, 2020, were included

DETAILED DESCRIPTION:
Data collection Data was collected deidentified admission from adult patients, with oxygen therapy. Data were extracted from clinical medical records and the electronic database of daily laboratory test results. Also, incomplete clinical records were included. The number of cases in the area during the study period determined the sample size, no formal hypotheses being implemented. All patients who met the inclusion criteria were included.

Study variables Demographic variables (sex and age), chronic medical histories (hypertension, diabetes and cancer), laboratory plasma, and serum-based biomarkers, as well as the mortality, mechanical ventilation, and length of stay, were considered. Leukocytosis was considered as a leucocyte count above 10 x 103/mcL, a cut point of INL> 10, d- dimer 500 U/L, DHL> 500U/L, low count of lymphocytes < 0·5103/mcL as risk factors exposure to death and mechanical ventilation.

A new variable was create combining the data of neutrophil count (ANC) and lymphocyte count (ALC) to obtain the neutrophil-to-lymphocyte ratio (NLR) (calculated dividing the ANC by the ALC).

Outcomes The hypothesis was formulated before the statistical analysis. Our primary outcomes were to 1) To describe the clinical characteristics of the Mexican population with SARS-CoV-2 infection, and 2) To determine the mortality risk factors in Covid-19.

Secondary outcomes included 1) To identify the chronic diseases related to Covid-19 in Mexican population and 2) To evaluate the differences in hematic and biochemical parameters between survivors and no survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥18 years)
2. Clinical (Positive RT-PCR for SARS-CoV-2 test) and radiological diagnosis of pulmonary infection by COVID-19
3. Diagnosis of acute respiratory distress syndrome clinical panel in accordance with Berlin 2012 criteria
4. Need of non-invasive ventilation (NIV or CPAP) or invasive ventilation (intubation)

Exclusion Criteria:

1. Previous diagnosis of severe liver or kidney failure.
2. Patients with Human Immunodeficiency Virus (HIV) infection.
3. Patients with previous hematological diseases (Leukemia) that condition alterations in blood counts.
4. Consumption of treatments with any type of immunosuppressants prior to admission that conditions low lymphocytes.
5. Patients with a diagnosis of active or non-active cancer.
6. Absence of a clinical record for monitoring the data.
7. Pregnancy.
8. Patients referred from other institutions for their medical care. Clinical records of patients who requested their voluntary discharge Clinical records that do not include information of the course of COVID-19 infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all hospitalized patients with the diagnosis of COVID-19 in the Hospital Regional de Alta Especialidad de Ixtapaluca (HRAEI) that were admitted in the Emergency ward, Intensive Care Unit (ICU) and all the reconversion areas.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Clinical complications and Mortality | 10 days
  To main aim of the study is to evaluate clinical complicatios and mortality in mexican Covid-19 patients
Neutrophil-Lymphocyte and Lymphocyte-Platelet ratio | 10 days
  To evaluate the association of the hematological ratios with the clinical complicatios and mortality in covid-19 patinets

OTHER OUTCOMES:
Hematic and biochemical parameters | 10 days
  To evaluate the differences in hematic and biochemical parameters between survivors and no survivors
Chronic diseases | 10 days
  To identify the chronic diseases in the patientss´medical records associated with the pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional de Alta Especialidad de Ixtapaluca, Ixtapaluca, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No